CLINICAL TRIAL: NCT02251626
Title: Assessing Bioavailability and Effects of Ubiquinol Supplementation on Biomarkers of Mitochondrial Function/Integrity, Metabolic Dysfunction, and Circulating Alarmins in Burn Patients
Brief Title: Assessing Bioavailability of CoQ10 Supplementation in Burn Patients
Acronym: CoQ10
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Principal Investigator, Masao Kaneki, Associate Professor/Associate Biochemist, Department of Anesthesia,Critical Care and Pain Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013P001111
Record Dates: First submitted 2014-09-20; First posted 2014-09-29 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Burn Injury
Keywords: MGH; Burn patient; Adult; CoQ10; Ubiquinol
MeSH Terms: conditions — Burns | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coenzyme Q10 (ubiquinol) (Experimental): Coenzyme Q10 (ubiquinol) group will be given 1,800 mg coenzyme Q10 (ubiquinol) per day
  Interventions: Dietary Supplement: coenzyme Q10
- Placebo for CoQ10 (ubiquinol) (Placebo Comparator): Placebo group will be given placebo only
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: coenzyme Q10 — It is a randomized and double blind study so patients or his/her doctor will not know which group s/he is in.
  Other Names: Ubiquinol supplement
  Arms: Coenzyme Q10 (ubiquinol)
Dietary Supplement: Placebo — It is a randomized and double blind study so patients or his/her doctor will not know which group s/he is in.
  Arms: Placebo for CoQ10 (ubiquinol)

SUMMARY:
To test the hypotheses that plasma and intracellular coenzyme Q10 levels will decline after burn injury and that ubiquinol supplementation will increase plasma and intracellular coenzyme Q10 levels in burn patients.

To test the hypothesis that ubiquinol supplementation ameliorates mitochondrial dysfunction/disintegrity and metabolic derangements, and decreases circulating alarmins (a.k.a. endogenous DAMPs) in burn patients as compared with placebo.

DETAILED DESCRIPTION:
Based on previous clinical studies and our preliminary preclinical data, we want to test the hypotheses that plasma and intracellular coenzyme Q10 levels are decreased after burn injury and that coenzyme Q10 (ubiquinol) supplementation reverses or ameliorates insulin resistance, metabolic derangements, mitochondrial dysfunction, and increased circulating DAMPs in burn patients. The aforementioned previous studies and preliminary data warrant a small-scale clinical study to evaluate coenzyme Q10 status, and bioavailability and efficacy of coenzyme Q10 (ubiquinol) supplementation in burn patients. Coenzyme Q10 (ubiquinol) supplementation could represent a novel, safe and low-cost strategy to improve the clinical outcome of burn patients. We are conducting a randomized, double-blind, placebo-controlled intervention study with anticipated enrollment of 50 subjects. Adult burn patients with 5% or greater of total body surface area (TBSA) burn at the Massachusetts General Hospital (MGH) Burn Center will be approached to consider study participation. All enrolled patients will be randomized to receive coenzyme Q10 (ubiquinol) supplementation or placebo. Blood samples will be used for evaluation of coenzyme Q10 concentration, mitochondrial DNA copy number, non-mitochondrial DAMPs (e.g., cell-free total DNA), and defective neutrophil migration.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 years and older, and below 85 yeas old
* Burn patients with 5% or greater of total body surface area burn
* Nutrition support: routine oral and/or enteral nutrition
* Enrolled within one week after burn injury
* Patient or guardian who is capable of giving full informed consent.
* Anticipated stay in the MGH Burn Unit: 5 days or more

Exclusion Criteria:

* < 5% TBSA burn
* Patients required full parenteral nutrition without oral or enteral nutrition support.
* Patients with liver disease (bilirubin greater than 3)
* Patients with thyroid disorders (thyroid disease which currently require treatment)
* Patients with malignancy under treatment
* Patients with mental illness who have impaired decision-making capacity (Mental illness defined by the presence of psychotropic medications and/or the diagnosis of psychiatric illness at the time of admission.) Patients with mental illness can be included unless it is determined by the psychiatrist covering the burn unit that they are unable to consent for themselves for other aspects of their care and treatment.)
* Patients with HIV*
* Pregnancy (as determined by routine admission labs)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Coenzyme Q10 Content in Peripheral Blood Mononuclear Cells | up to four weeks
Plasma Coenzyme Q10 Concentration | up to four weeks

SECONDARY OUTCOMES:
Plasma Mitochondrial DNA Concentration | up to four weeks
Plasma cytokine concentrations | up to four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masao Kaneki, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No